CLINICAL TRIAL: NCT06522568
Title: Toward Optimization of a Mammography Decision Aid and Clinician Communication Intervention Trial for Rural Settings
Brief Title: Testing a Mammography Decision Intervention in a Rural Setting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, Mark A. Creager, Professor of Medicine, Geisel School of Medicine, Dartmouth; Professor of Surgery, Geisel School of Medicine, Dartmouth, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY02002381
Record Dates: First submitted 2024-07-17; First posted 2024-07-26 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Screening
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual Care (No Intervention): Usual care.
- MyMammogram (Experimental): Patient uses MyMammogram prior to appointment.
  Interventions: Behavioral: MyMammogram
- MyMammogram plus provider communication (Experimental): Patient uses MyMammogram prior to appointment. Provider receives a summary from MyMammogram prior to appointment.
  Interventions: Behavioral: MyMammogram; Other: Provider communication

INTERVENTIONS:
Behavioral: MyMammogram — An online breast cancer screening decision aid
  Arms: MyMammogram; MyMammogram plus provider communication
Other: Provider communication — Provider will be provided with information from MyMammogram that includes patient's breast cancer risk and preferences for mammograms prior to the appointment
  Arms: MyMammogram plus provider communication

SUMMARY:
The overall objective of this COBRE pilot project is to enhance the design of a 3-arm cluster randomized trial that will test the efficacy and mechanism of effect of the MyMammogram DA with or without a provider communication intervention. This will be accomplished through two aims: (1) Refine, with community partner input, a clinical trial protocol to optimize engagement among patients and primary care providers (PCPs) practicing in rural settings. In consultation with patients, PCPs, and informatics experts, the study team will refine site selection, randomization, patient and PCP recruitment, and data collection protocols to meet the needs of the rural health care delivery system and participants. The result of this aim will be a modified protocol and intervention strategy that is acceptable to partners. (2) Adapt and test trial and intervention implementation features to achieve protocol acceptance and adherence. The investigators will pilot the adapted three-arm randomized trial protocol in rural primary care settings that compares the MyMammogram DA with or without a risk summary provided to the PCP pre-visit, relative to usual care. Implementing the trial in two phases (n=15 each) will systematically identify barriers and facilitators to trial participation to refine protocols. Participants will receive acceptability surveys and investigators will conduct qualitative interviews with patients and PCPs to understand experiences with trial implementation from multiple perspectives.

DETAILED DESCRIPTION:
This is a three-arm randomized pilot trial that will enroll 30 participants over two study phases. The main objective is to achieve data on trial feasibility (recruitment, retention, randomization, adherence, and acceptability). The primary outcome is Intervention Acceptability.

Procedures: PCPs will be randomized to one of the three arms to prevent contamination across patients (usual care, decision aid, decision aid + clinician communication). Patients will be considered for enrollment if they are aged 40-49, English or Spanish-speaking, have an upcoming primary care visit within 4 weeks, no history of breast cancer, ductal carcinoma in situ, lobular carcinoma in situ, or atypical hyperplasia, and no mammogram within the past 12 months. These patients will be identified via the electronic health record using routine data reports provided to the study team.

Data Collection: Surveys will be conducted at baseline (pre-intervention), post-DA and Post-Visit. Mammography screening information will be collected via medical records, and implementation data will be completed with patients and clinicians who were exposed to the decision aid intervention.

Analysis: All feasibility metrics will be summarized quantitatively, distributions examined for central tendency and spread, and all data assessed for completeness. Data will be presented in a tabular format, with means and standard deviations summarized for the Acceptability of Intervention Measure. Process data will likewise be summarized, reporting proportions of participants meeting each metric (recruitment, retention, randomization, adherence).

ELIGIBILITY:
Patient Inclusion Criteria:

* Females
* Aged 39-49
* Upcoming appointment with a participating primary care provider (within 4 weeks)
* English or Spanish-speaking

Patient Exclusion Criteria:

* Personal history of breast cancer (including lobular carcinoma in situ and ductal carcinoma in situ or atypical hyperplasia)
* Mammogram in the prior 12 months

Clinician inclusion: Any practicing primary care provider at a participating site.

Ages: 39 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Intervention acceptability | within one day of completing the intervention
  The acceptability e-scale is a 6-item measure for electronically-delivered interventions, where higher scores indicate greater acceptability. Scores range from 6-30.

SECONDARY OUTCOMES:
Recruitment feasibility | 4 weeks
  Measured as the proportion of eligible participants who receive an initial outreach letter and complete the consent process and enroll prior to their clinical visit.
Retention feasibility | 8 weeks
  Proportion of participants enrolled who complete all study survey time points, reported per trial arm

OTHER OUTCOMES:
Knowledge | enrollment and within one day of completing the intervention
  10-item measure of breast cancer and screening knowledge that is summed for a score from 0-10 (0 indicates lower knowledge, 10 indicates higher knowledge).
Decisional Quality | enrollment, within one day of completing the intervention, within one day of completing a clinical visit
  Decisional Quality is measured using the Decisional Conflict Scale for Low Literacy, a 10-item measure. Scores Range 0-100. Lower scores indicate better decisional quality (lower conflict).
Screening Intentions | enrollment, within one day of completing the intervention, within one day of completing a clinical visit
  Screening intentions are using two methods. 1) As the likelihood of obtaining a mammogram in the next year (5-point Likert scale); and 2) Using 2 items to measure age at which someone intends to begin screening (40, 45, 50, other) and interval (annual, biennial, other).
Shared Decision-Making | within one day of completing a clinical visit
  Shared Decision Making will be assessed with the 3-item, validated CollaboRATE measure. Scored 0-100 (higher scores indicate more shared decision-making).
Self-efficacy | enrollment and within one day of completing a clinical visit
  Measured using a validated scale measuring perceived confidence one's personal ability to obtain a mammogram. Ten items are summed, with a theoretical score range from 5-10 (higher scores indicate better self-efficacy).

CONTACTS AND LOCATIONS:
Locations (1):
- Cheshire Medical Center, Keene, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No